CLINICAL TRIAL: NCT03174509
Title: Is Positive Pressure Extubation Safe Procedure? A Randomized Non-inferiority Trial.
Brief Title: Is Positive Pressure Extubation a Safe Procedure?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Donación Francisco Santojanni (Other)
Responsible Party: Principal Investigator, Mauro Andreu, Physical Therapist, Hospital Donación Francisco Santojanni
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGADFS14012016-01
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Complication
Keywords: airway extubation; positive-pressure respiration; suction; ventilator weaning

STUDY DESIGN:
Intervention Model Description: Non-inferiority trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The pre and post extubation parameters are recorded by an outcome assessor who do not know the assigned extubation method.
  The assigned extubation method is coded to minimize potential bias during data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Pressure Extubation (Active Comparator): Positive pressure extubation is used for patients in this group.
  Interventions: Procedure: Positive pressure extubation
- Traditional Extubation (Active Comparator): Traditional extubation is used for patients in this group.
  Interventions: Procedure: Traditional during extubation

INTERVENTIONS:
Procedure: Positive pressure extubation — Positive pressure ventilation without endotracheal aspiration/suction during extubation procedure.
  Arms: Positive Pressure Extubation
Procedure: Traditional during extubation — Spontaneous ventilation with endotracheal aspiration/suction during extubation procedure.
  Arms: Traditional Extubation

SUMMARY:
Laboratory studies suggest extubation with positive pressure because it reduces the volume of secretions filtered into the distal airway. The aim of this non inferiority study is to evaluate the safety of the extubation technique under positive pressure with respect to the traditional technique (with suction and without positive pressure in the airways).

DETAILED DESCRIPTION:
The extubation procedure consists of the removal of the endotracheal tube when it is no longer required. The literature reports two methods of extubation: the named traditional method (with suction and without positive pressure in the airways) and the positive pressure method. Laboratory studies suggest extubation at positive pressure because it reduces the volume of secretions filtered into the distal airway. Prior to apply it into clinical practice the investigators of this study consider is a priority to guarantee the safety of the positive pressure extubation method in terms of presence of complications.

The aim of this non-inferiority study is to compare the incidence of complications between both extubation techniques in adult patients with invasive mechanical ventilation.

The hypothesis of this study is that applying positive pressure during cuff deflation and extubation is not inferior to the traditional method in the incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Invasive Mechanical Ventilation with endotracheal tube.
* 18 years and older.
* Successful 30 minutes spontaneous breathing trial (SBT).
* Extubation Criteria.
* Informed consent.

Exclusion Criteria:

* Previous airway surgery or injury.
* Non-Invasive Ventilation as weaning method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence/A presence/absence of complications after extubation | 60 minutes
  Clinical Evidence of at least one of the next complications: persistent cough, airway obstruction, post-obstructive pulmonary edema, bronchospasm, desaturation, vomiting, tachycardia, arterial hypertension.

SECONDARY OUTCOMES:
Pneumonia | 72 hours
  Presence of fever, leukocytosis, purulent secretions and a new pulmonary infiltrate on chest radiography
Reintubation | 72 hours
  Intubation requirement after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Mauro F Andreu, PT, Principal Investigator — Hospital D. F. Santojanni
Locations (1):
- Hospital Santojanni, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andreu MF, Salvati IG, Donnianni MC, Ibanez B, Cotignola M, Bezzi M. Effect of applying positive pressure with or without endotracheal suctioning during extubation: a laboratory study. Respir Care. 2014 Dec;59(12):1905-11. doi: 10.4187/respcare.03121. Epub 2014 Nov 25. PMID 25425709
- [Derived] Andreu MF, Dotta ME, Bezzi MG, Borello S, Cardoso GP, Dib PC, Garcia Schustereder SL, Galloli AM, Castro DR, Di Giorgio VL, Villalba FJ, Bertozzi MN, Carballo JM, Martin MC, Brovia CC, Pita MC, Pedace MP, De Benedetto MF, Delli Carpini J, Aguirre P, Montero G. Safety of Positive Pressure Extubation Technique. Respir Care. 2019 Aug;64(8):899-907. doi: 10.4187/respcare.06541. Epub 2019 Mar 26. PMID 30914493